CLINICAL TRIAL: NCT07287592
Title: Glutamine for the Prophylaxis of Vincristine-induced Neuropathy in Children and Adolescents With Cancer. A Single Center Study
Brief Title: Glutamine for the Prophylaxis of Vincristine-induced Neuropathy in Children and Adolescents With Cancer.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU R 146/2021
Record Dates: First submitted 2025-11-30; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Neuropathy; Cancer
Keywords: vincristine; cancer; neuropathy
MeSH Terms: conditions — Neoplasms | interventions — Glutamine

STUDY DESIGN:
Intervention Model Description: A block-randomization scheme will be generated by computer software. Patients fulfilling the inclusion criteria will then be randomly distributed between glutamine and the standard of care therapy in a 1:1 ratio.
  * Intervention arm: Thirty five patients will receive glutamine in a dose of 6 g /m2 twice daily (up to a maximum of 10 g/dose) for forteen consecutive days starting from induction and forteen days starting from continuation . The dose used in the current study is determined by prior adult studies described a significant beneficial effect of glutamine on oxaliplatin and paclitaxel-induced peripheral neuropathy (Wang et al., 2007)
  * Standard of care arm: Thirty five patients will be assigned as a control group with no medication given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Active Comparator): Thirty five patients will receive glutamine in a dose of 6 g /m2 twice daily (up to a maximum of 10 g/dose) for forteen consecutive days starting from induction and forteen days starting from d1 of continuation . The dose used in the current study is determined by prior adult studies described a significant beneficial effect of glutamine on oxaliplatin and paclitaxel-induced peripheral neuropathy (Wang et al., 2007)
  Interventions: Drug: Glutamine (Pharmacological doses)
- Standard of care arm (No Intervention): the usual standard of care

INTERVENTIONS:
Drug: Glutamine (Pharmacological doses) — glutamine is an essential amino acid. It will be provided in a powder form. It will be dissolved in at least 8 ounces of hot or cold liquid. It can also be mixed with a soft food such as pudding
  Arms: Intervention arm

SUMMARY:
The goal of this clinical trial is to assess the efficacy of glutamine in preventing the occurrence of vincristine induced neuropathy and to compare the reduction in rate of any dose reductions and premature chemotherapy discontinuation rates due to peripheral neuropathy between those who treated with glutamine and those who did not.

Participants will:

receive glutamine in a dose of 6 g /m2 twice daily (up to a maximum of 10 g/dose) for 14 consecutive days from d 1 of induction and 14 days from d1 of continuation .

• Subjects will be asked to return for a complete study assessments visit every 14-days during supplementation period for a total of 4 visits Keep a diary of their symptoms of neuropathy and compliance to treatment and any adverse event

ELIGIBILITY:
Inclusion Criteria:

1. No sex predilection.
2. Age: 6 years to 18 years
3. Children and adolescents diagnosed with hematological malignancy or solid tumors expected to receive a cumulative dose of 6 mg/m2 of VCR over a 12 week period (or >6 mg/m2 if individual VCR doses were capped at 2 mg) according to their primary cancer treatment protocol
4. Patients with score less than 5 on pediatric modified total neuropathy scale at Time 0

Exclusion Criteria:

1. Patients with CNS tumors
2. Patients with focal neurologic findings or CNS metastasis Patients with premorbid developmental disorders, neuromuscular disorders or diabetes mellitus Patients with recurrent disease already exposed to >8 mg/m2 of VCR Patients with score more than 5 on pediatric modified total neuropathy scale

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
safety outcome | 12 months
  The primary safety endpoint was the the number of participants who will report bleeding tendency episodes and number of participants with significant impairment of liver or kidney functions
primary objective outcome | 3 months
  the number of participants who develop neuropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No